CLINICAL TRIAL: NCT01864291
Title: Study of the Nucleus 24 and ABI541 Auditory Brainstem Implants in Pediatric Non-Neurofibromatosis Type 2
Brief Title: Auditory Brainstem Implant (ABI) in Pediatric Non-Neurofibromatosis Type 2 Subjects
Acronym: ABI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by IRB
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Dr. Daniel Lee, Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-028H
Record Dates: First submitted 2013-05-22; First posted 2013-05-29 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Bilateral Hearing Loss for Causes Other Than Tumors
Keywords: Auditory Brainstem Implant; ABI; Nucleus 24; Deafness; Hearing loss; Non-tumor; Non-NF2; Pediatric; ABI541
MeSH Terms: conditions — Deafness; Hearing Loss | interventions — Ankle Brachial Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Non-NF2 ABI surgery (Experimental): All subjects will be part of a single arm involving placement of the ABI541 Auditory Brainstem Implant (ABI) device. The Nucleus 24 was discontinued and is no longer available.
  Interventions: Device: Nucleus 24 (discontinued) and ABI541 Auditory Brainstem Implants (ABI)

INTERVENTIONS:
Device: Nucleus 24 (discontinued) and ABI541 Auditory Brainstem Implants (ABI) — Nucleus ABI541 Auditory Brainstem Implant (ABI) surgery followed by device activation, testing, and clinical assessment for five years following surgery.
  Other Names: ABI, Nucleus 24, ABI541, Nucleus Profile, Cochlear Americas

SUMMARY:
The purpose of this research study is to determine whether Auditory Brainstem Implant (ABI) can improve hearing in children who are deaf and cannot receive a cochlear implants.

DETAILED DESCRIPTION:
The goal of this MEEI Auditory Brainstem Implant (ABI) research study is to find new ways to improve hearing in children who are deaf and cannot receive a cochlear implant. The ABI is a surgically placed bionic implant that converts sounds into electrical signals that are directly transmitted to the cochlear nucleus, the first auditory center of the brain. For many years, ABIs have improved the hearing of patients who are deaf due to brain tumors associated with a genetic syndrome called Neurofibromatosis Type 2 (NF2). However, a number of recent studies suggest that deaf patients who do not have NF2 and are not eligible for a cochlear implant may also benefit from placement of an ABI. These preliminary studies suggest that these non-NF2 or "nontumor" patients may actually have better outcomes after ABI surgery than patients suffering from NF2. Children appear to be particularly good candidates because of their developmental plasticity and in many studies, outcomes are more favorable in children that adults. Patients who do not have NF2 and are deaf due to abnormalities in their hearing nerves or inner ears from congenital malformations, infection, disease, or injury are not cochlear implant candidates and there are no other options to improve hearing in these cases except for the ABI. Thus, the purpose of our study is to carefully analyze whether ABI surgery improves the hearing and quality of life of non-NF2 children based on subjective and objective measures of their hearing before and after ABI surgery. In particular, we plan to study ABI outcomes in non-NF2 pediatric patients, characterize the parameters used on their devices, and determine the safety profile of ABIs in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-linguistic hearing loss (birth-5 yrs.; age at ABI implantation 18 months-5yrs) with both:

   1. MRI +/- CT evidence of one of the following:

      * Cochlear nerve deficiency
      * Cochlear aplasia or severe hypoplasia
      * Severe inner ear malformation
      * Post-meningitis ossification
   2. When a cochlea is present or patent with a normally appearing cochlear nerve, lack of significant benefit from CI despite consistent use (>6 mo.)

      * No or limited speech perception ability (limited to pattern perception on closed set testing materials using the CI)
      * Lack of progress in auditory skills development
2. Post-linguistic hearing loss (<18 yrs. of age) with both:

   1. Loss or lack of benefit from appropriate CI without the possibility for revision or contralateral implantation. Examples might include:

      * Post-meningitis ossification
      * Bilateral temporal bone fractures with cochlear nerve avulsion
      * Failed revision CI without benefit
   2. Previously developed open set speech perception and auditory-oral language skills
3. No medical contraindications
4. Willing to receive the appropriate meningitis vaccinations
5. No or limited cognitive/developmental delays which would be expected to interfere with the child's ability to cooperate in testing and/or programming of the device, in developing speech and oral language, or which would make an implant and subsequent emphasis on aural/oral communication not in the child's best interest
6. Strong family support including language proficiency of the parent(s) in the child's primary mode of communication as well as written and spoken English.
7. Reasonable expectations from parents including a thorough understanding:

   * of potential benefits and limitations of ABI
   * of parental role in rehabilitation
   * that the child may not develop spoken language as a primary communication mode or even sufficient spoken language to make significant academic progress in an aural/oral environment
8. Involvement in an educational program that emphasizes development of auditory skills with or without the use of supplementary visual communication.
9. Able to comply with study requirements including travel to investigation sites and clinic visits.
10. Informed consent for the procedure from the child's parents.

Exclusion Criteria:

1. Pre- or post-linguistic child currently making significant progress with CI - This will be considered if a child is progressing along the expected speech reception hierarchy (SRI-Q) as detailed by Wang et al (50). Even for the very young children (18 months of age with 6 months of use), nearly all children with a good auditory signal from their CI will have reached ceiling effects on the IT-MAIS and have pattern perception beyond chance using the ESP (50). Moreover, there will evidence of improvement in these metrics over time.
2. MRI evidence of one of the following:

   * normal cochlea and cochlear nerves or NF2
   * brainstem or cortical anomaly that makes implantation unfeasible
3. Clear surgical reason for poor CI performance that can be remediated with revision CI or contralateral surgery rather than ABI.
4. Intractable seizures or progressive, deteriorating neurological disorder
5. Unable to participate in behavioral testing and mapping with their CI. If this appears to be an age effect, ABI will be delayed until we can be assured that the child will be able to participate, as reliable objective measures of mapping are currently not available for mapping these devices.
6. Lack of potential for spoken language development. This will be considered the case when evidence of the following exist:

   * Severe psychomotor retardation, autism, cerebral palsy, or developmental delays beyond speech that would preclude usage of the device and oral educational development. Autism is a special case where there is the potential for delayed presentation. When early signs are considered present, we will request a comprehensive developmental assessment for further evaluation prior to considering routine evaluation.
7. Unable to tolerate general anesthesia (cardiac, pulmonary, bleeding diathesis, etc.).
8. Need for brainstem irradiation
9. Unrealistic expectations on the part of the subject/family regarding the possible benefits, risks and limitations that are inherent to the procedure and prosthetic device.
10. Unwilling to sign the informed consent.
11. Unwilling to make necessary follow-up appointments.

Ages: 18 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Lee, MD FACS, Principal Investigator — MEEI/MGH
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colletti V, Shannon RV, Carner M, Veronese S, Colletti L. Complications in auditory brainstem implant surgery in adults and children. Otol Neurotol. 2010 Jun;31(4):558-64. doi: 10.1097/MAO.0b013e3181db7055. PMID 20393378
- [Background] Sennaroglu L, Ziyal I, Atas A, Sennaroglu G, Yucel E, Sevinc S, Ekin MC, Sarac S, Atay G, Ozgen B, Ozcan OE, Belgin E, Colletti V, Turan E. Preliminary results of auditory brainstem implantation in prelingually deaf children with inner ear malformations including severe stenosis of the cochlear aperture and aplasia of the cochlear nerve. Otol Neurotol. 2009 Sep;30(6):708-15. doi: 10.1097/MAO.0b013e3181b07d41. PMID 19704357
- [Background] Choi JY, Song MH, Jeon JH, Lee WS, Chang JW. Early surgical results of auditory brainstem implantation in nontumor patients. Laryngoscope. 2011 Dec;121(12):2610-8. doi: 10.1002/lary.22137. PMID 22109761
- [Background] Colletti V, Shannon R, Carner M, Veronese S, Colletti L. Outcomes in nontumor adults fitted with the auditory brainstem implant: 10 years' experience. Otol Neurotol. 2009 Aug;30(5):614-8. doi: 10.1097/MAO.0b013e3181a864f2. PMID 19546832
- [Background] Colletti V, Carner M, Miorelli V, Guida M, Colletti L, Fiorino F. Auditory brainstem implant (ABI): new frontiers in adults and children. Otolaryngol Head Neck Surg. 2005 Jul;133(1):126-38. doi: 10.1016/j.otohns.2005.03.022. PMID 16025066
- [Background] Colletti V. Auditory outcomes in tumor vs. nontumor patients fitted with auditory brainstem implants. Adv Otorhinolaryngol. 2006;64:167-185. doi: 10.1159/000094651. PMID 16891842
- [Background] Colletti L, Zoccante L. Nonverbal cognitive abilities and auditory performance in children fitted with auditory brainstem implants: preliminary report. Laryngoscope. 2008 Aug;118(8):1443-8. doi: 10.1097/MLG.0b013e318173a011. PMID 18496153

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-NF2 ABI Surgery: Implantation with Auditory Brainstem Implant (ABI) device and clinical follow-up
Period: Overall Study
Arm/Group | Non-NF2 ABI Surgery
Started | 9
Completed | 7 (7/9 subjects had a minimum of one year followup since enrollment.)
Not Completed | 2
Not completed — need for revision surgery | 2

BASELINE CHARACTERISTICS:
Arm/Group | Non-NF2 ABI Surgery
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: months] | 27 [15 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9
Sound detection via pure-tone threshold audiometry [Mean (Full Range); unit: dB HL] — As all participants have (1) absent cochleae or absent cochlear nerves or (2) anatomic conditions of the inner ear that preclude the use of a traditional cochlear implant array, it was expected that participants would have profound hearing loss at baseline and no residual hearing. Therefore, it was hypothesized that sound detection would be at the upper limit of clinical testing.
  The decibel unit is plotted on a logarithmic scale; higher values represents worse hearing. 120 dB HL represents the upper limit of clinical testing.
  dB HL | 120 [120 to 120]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major or Minor ABI Complications
Description: We will track any major and minor complications peri-operatively and post-operatively in all study participants. Major complications include mortality, cerebellar contusion, facial palsy, meningitis, lower cranial neuropathy, hydrocephalus, pseudomeningocele and CSF leak. Minor complications include transient hydrocephalus, wound seroma, minor infections, balance problems, transient nerve palsies, transient dysphonia or difficulty swallowing, headache, flap problems, and non-auditory side effects. These complications will be tracked through serial clinical exams as well as patient recorded questionnaires to determine the safety profile of ABI surgery.
Time Frame: 1 year from date of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Non-NF2 ABI Surgery
Number analyzed (Participants) | 9
Participants
  Major Complications | 2
  Minor Complications | 7

2. Secondary Outcome: Change in Pure Tone Threshold (dB HL) Using the ABI
Description: We will complete audiometric threshold testing and speech based tests to determine performance before and after ABI surgery.
  The measure data value was calculated as mean threshold shift in dB HL from pre-surgery (or baseline) to postoperatively (following activation of the ABI) across subjects analyzed. Only those subjects that had auditory perception abilities were included. 2/9 subjects did not have auditory perception and are not using their devices.
  The outcome measure time frame varies across subjects based on available followup data as this study was stopped early.
  Audiometric testing will include:
  • Behavioral pure tone threshold average (PTA) in both aided (with ABI) and unaided (without ABI)
Time Frame: 1-4 years from date of surgery
Population: 2/9 subjects required revision surgery for device issues and were not included in this analysis as they did not complete the study. An additional 2/9 subjects did not have auditory perception and are not using their device and were also not included in this analysis.
Measure: Mean (Full Range); unit: dB HL
Arm/Group | Non-NF2 ABI Surgery
Number analyzed (Participants) | 5
dB HL | 73 [65 to 85]

3. Secondary Outcome: Number of Participants With Similar eABR Morphology on the Day of ABI Activation Compared to Intraoperative Responses
Description: We will measure and record the specific programmed parameters of the ABI device. Intraoperatively, evoked Auditory Brainstem Response (eABRs) will be recorded and saved. These tracings and data will be compared to the settings on activation to determine whether the same electrodes are appropriately positioned. By following these measures, we will be able to capture how electrophysiologic parameters vary (if at all) over time.
  The outcome measure data are the number of subjects whose eABR morphology was similar on the day of activation (4 to 8 weeks following surgery) as recorded intraoperatively during ABI surgery.
Time Frame: 4 to 8 weeks after surgery (day of activation under anesthesia)
Measure: Count of Participants; unit: Participants
Arm/Group | Non-NF2 ABI Surgery
Number analyzed (Participants) | 9
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 5 years post-operatively for purposes of the study, though all participants have ongoing routine safety monitoring as part of their clinical care.
Arm/Group | Non-NF2 ABI Surgery
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 7/9
Other Adverse Events (participants affected / at risk) | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-NF2 ABI Surgery (N=9)
device failure (Product Issues) | 3 (3)
no auditory perception (Product Issues) | 2 (2) — no auditory perception at awake activation
nausea and vomiting (Gastrointestinal disorders) | 2 (2) — admitted to hospital for management of symptoms
oxygen desaturation (Respiratory, thoracic and mediastinal disorders) | 2 (2) — oxygen desaturation in PICU treated with steroids, one case associated with reactive airway disease
upper respiratory infection with shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-NF2 ABI Surgery (N=9)
ear infection (Ear and labyrinth disorders) | 2 (2)
anemia (Blood and lymphatic system disorders) | 1 (1) — incidental finding per pre-op labs
post-intubation airway edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
blister (Skin and subcutaneous tissue disorders) | 1 (1) — 2-3cm right heel blister
abcess (Skin and subcutaneous tissue disorders) | 1 (1) — stitch abcess
swelling after fall (General disorders) | 1 (1) — fell out of crib, developed swelling that later resolved
pain (General disorders) | 1 (1) — post-surgical pain
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
postoperative edema (General disorders) | 1 (1) — Fluid accumulation around incision site
bradycardia (Cardiac disorders) | 1 (1)
bruxism (General disorders) | 1 (1) — increase in grinding teeth while using the device
ear drainage (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT01864291/Prot_SAP_000.pdf